CLINICAL TRIAL: NCT01619137
Title: Comparison of the Effect of Water and Soap Irrigation With With Povidone-iodine And Normal Salin Treatment of Patients With Ununion Laparatomy or Episiotomy Wound ( a Pilot Study)
Brief Title: Soap Versus Normal Salin Plus Povidone-iodine in Ununion Wound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aida Najafian (Other)
Responsible Party: Sponsor-Investigator, Aida Najafian, Specialist, Hormozgan University of Medical Sciences
Organization: Hormozgan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: soap in ununion wound
Record Dates: First submitted 2012-01-19; First posted 2012-06-14 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Wound
Keywords: ununion wound; soap; irrigation; Povidone-iodine; normal salin
MeSH Terms: conditions — Wounds and Injuries | interventions — Water; Soaps; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Povidone-iodine And normal salin (Active Comparator): 40 patients with complaint of ununion wound of laparatomy or episiotomy coming to Gynecologist's office or hospital enrolled to this study randomly recieve Povidone-iodine And normal salin treatment.
  Interventions: Drug: Povidone-iodine And normal salin treatment
- water and soap (Active Comparator): 40 patients coming to Gynecologist's offices or hospital with complaint of ununion wound of laparatomy or episiotomy in Bandarabbas enrolled to this study and randomly recieve water and soap to irrigation of the wound (it's not require to be at hospital), washing is for each 6-8 hours per day. and if not difference seen after 4 day, treatment change to Povidone-iodine And normal salin.
  Interventions: Drug: water and soap

INTERVENTIONS:
Drug: water and soap — water and soap for 6-8 hours per day.
  Arms: water and soap
Drug: Povidone-iodine And normal salin treatment — use of Povidone-iodine And normal salin treatment for irrigation of ununion laparatomy or episiotomy wound.
  Arms: Povidone-iodine And normal salin

SUMMARY:
Comparison of the effect of water and soap irrigation with Povidone-iodine And normal salin treatment of patients with ununion laparatomy or episiotomy wound ( a pilot study)

DETAILED DESCRIPTION:
IN Comparison of the effect of water and soap irrigation with Povidone-iodine And normal salin treatment of patients with ununion laparatomy or episiotomy wound ( a pilot study), We use soap in one group and Povidone-iodine And normal salin in other group for irrigation of ununion laparatomy or episiotomy wound.it's require the patients in Povidone-iodine And normal salin group be at hospital till wound be able to closed.

ELIGIBILITY:
Inclusion Criteria:

* all the women coming to Shariati hospital or Gynecologist's office with complain of ununion wound of laparatomy or episiotomy enroll to this study

Exclusion Criteria:

* patients not satisfacted to participant in the study exclude of it

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
number of admission day | 1 month
  number of days the patients in each group admitted in hospital

SECONDARY OUTCOMES:
complication of each treatment | 1 months
  complications include of : infection, reopening of wound, and measurment of opening of wound.

CONTACTS AND LOCATIONS:
Overall Officials: Aida Najafian, Principal Investigator — Hormozgan University of Medical Science (HUMS)
Locations (1):
- Bandarabbas, Bandarabbas, Hormozgan, Iran